CLINICAL TRIAL: NCT01255254
Title: The Effect of Oral Hygiene and Full Mouth Scaling on Metabolic Control in Patients With Type II Diabetes
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Department of Periodontology, School of Gradute Dentistry Rambam Health care campus Haifa, Israel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RMB 0350-10 CTIL
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-08

CONDITIONS: Gingival Scaling; Metabolic Control
Keywords: he effect of gingival scaling on Metabolic control

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Scaling group (Experimental): The experimental group will receive oral hygiene instruction (OHI) and full-mouth scaling using standard rigid Gracey curettes (Hu-Friedy® Manufacturing Inc., Chicago, IL, USA) and ultrasonic instrumentation (EMS piezoelectric system, Electro Medical Systems, Nyon, Switzerland) at week 1-2 and at a second reinforcement visit at 6-8 weeks. Subjects will also be instructed to rinse with 10ml of Chlorhexidine 0.2% mouthrinse twice daily for 30 seconds for the duration of the study.
  Interventions: Procedure: Gingival scaling
- B: Control group (No Intervention): The control group will receive no periodontal treatment during the study. After completion of the study, these patients will be given oral hygiene instruction and a full mouth scaling.

INTERVENTIONS:
Procedure: Gingival scaling — Oral hygeine instruction and gingival scaling using hand and ultrsonic instruments.
  Arms: A: Scaling group

SUMMARY:
The aim of the study is to evaluate the effect of non-surgical periodontal therapy, consisting of oral hygiene instruction, full mouth scaling and an antimicrobial rinse on the metabolic control of chronic periodontitis patients with type II diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25- 75 years;
2. Type 2 diabetes;
3. Chronic periodontitis with 2 or more teeth with CAL≥6mm and one site with a PD≥5mm ("established periodontitis")16

Exclusion Criteria:

1. Periodontal treatment within the last 3 months
2. The use of antibiotics within the last 4 weeks
3. Pregnancy or the intention to be pregnant in the next 4 months

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Metabolic control | 3 months
  Blood sample that measures fasting plasma glucose and the HbA1c level.

SECONDARY OUTCOMES:
Inflammation | 3 months
  Blood sample to measure C reactive protein (inflammatory marker).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology, School of Graduate Dentistry Rambam Health care campus, Haifa, Israel